CLINICAL TRIAL: NCT01600222
Title: A Phase 2 Maximal Use Systemic Exposure (MUSE) Study Evaluating the Safety and Efficacy of LEO 90100 Used Once Daily in Subjects With Extensive Psoriasis Vulgaris
Brief Title: Effect of LEO 90100 on the HPA Axis and Calcium Metabolism in Subjects With Extensive Psoriasis VulgarisExtensive Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEO 90100-30
Record Dates: First submitted 2012-05-08; First posted 2012-05-17 (Estimated); Results first posted 2016-09-16 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2016-07

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEO 90100 (Experimental)
  Interventions: Drug: LEO 90100

INTERVENTIONS:
Drug: LEO 90100 — Calcipotriol 50 mcg/g (as hydrate) and betamethasone 0.5 mg/g (as dipropionate)

SUMMARY:
A Phase 2 Maximal Use Systemic Exposure (MUSE) study evaluating the safety and efficacy of LEO 90100 used once daily in subjects with extensive psoriasis vulgaris.

DETAILED DESCRIPTION:
The purpose of the present study is to assess the systemic safety of LEO 90100. Although LEO 90100 contains the same active ingredients in the same concentration as DAIVOBET/DOVOBET/TACLONEX ointment, the degree of absorption of the active ingredients from the new formulation may differ. Systemic safety will be assessed through the effect of LEO 90100 on calcium metabolism and HPA axis function under maximum use conditions (i.e., in subjects with very extensive psoriasis on the trunk, limbs and scalp, using up to 120g per week of LEO 90100 for up to 4 weeks). Data from this study, together with the measurements of albumin-corrected serum calcium and the calcium:creatinine ratio in spot urine samples in the planned phase 2 and 3 studies in the development program for LEO 90100, are expected to provide adequate information with respect to the systemic safety of LEO 90100.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained prior to any trial related activities (including any washout period)
* Age 18 years or above
* Either sex
* Any race or ethnicity
* Any skin type
* Attending a hospital out-patient clinic or the private practice of a dermatologist for treatment of psoriasis vulgaris
* At SV2 and Day 0 (Visit 1), a clinical diagnosis of psoriasis vulgaris of at least 6 months duration involving the trunk and/or limbs and the scalp which is;

  * amenable to topical treatment with a maximum of 120g of study medication per week
  * of an extent of between 15 and 30% of the body surface area (BSA) excluding psoriatic lesions of the face, genitals and skin folds
  * including at least 30% scalp involvement
  * of at least a moderate disease severity according to the investigators global assessment (IGA)
* At SV2, a normal HPA axis function including a serum cortisol concentration above 5 mcg/dl before ACTH-challenge and above 18 mcg/dl 30 minutes after ACTH-challenge
* At SV2, an albumin-corrected serum calcium below the upper reference range limit
* At SV2, females of child-bearing potential must have a negative urine pregnancy result
* Females of child-bearing potential must agree to use a highly effective method of contraception during the study. A highly effective method of birth control is defined as one which results in a low failure rate (less than 1% per year)
* Able to communicate with the investigator and understand and comply with the requirements of the study

Exclusion Criteria:

* A history of allergic asthma, serious allergy or serious allergic skin rash
* Known or suspected hypersensitivity to component(s) of LEO 90100 or CORTROSYN (including cosyntropin/tetracosactide)
* Systemic treatment with corticosteroids (including inhaled and nasal steroids) within 12 weeks prior to SV2
* Systemic treatment with biological therapies (whether marketed or not marketed), with a possible effect on psoriasis vulgaris within the following time period prior to Day 0 (Visit 1);

  * etanercept - within 4 weeks
  * adalimumab, alefacept, infliximab - within 8 weeks
  * ustekinumab - within 16 weeks
  * other products - within 4 weeks/5 half-lives (whichever is longer)
* Subjects who have received treatment with any non-marketed drug substance (i.e. a drug which has not yet been made available for clinical use following registration) within 4 weeks/5 half-lives (whichever is longer) prior to Day 0 (Visit 1)
* Systemic treatment with all other therapies with a possible effect on psoriasis vulgaris (e.g. retinoids, methotrexate, cyclosporine and other immunosuppressants) within 4 weeks prior to Day 0 (Visit 1)
* PUVA therapy within 4 weeks prior to Day 0 (Visit 1)
* UVB therapy within 2 weeks prior to day 0 (Visit 1).
* Topical treatment with corticosteroids or vitamin D analogues on any body location within 2 weeks prior to SV2
* Any topical treatment of psoriasis vulgaris on the trunk, limbs or scalp (except for emollients and non-medicated shampoos) within 2 weeks prior to Day 0 (Visit 1)
* Planned initiation of, or changes to, concomitant medication that could affect psoriasis vulgaris (e.g., betablockers, antimalarials, lithium, ACE inhibitors) during the study
* Oral calcium supplements, vitamin D supplements, bisphosphonates or calcitonin within 4 weeks prior to SV2. Note: Stable doses of oral vitamin D supplementation ≤400 IU/day is permitted provided there are no dose adjustments during the study period
* Planned initiation of, or changes to concomitant medication that could affect calcium metabolism (e.g. antacids, thiazide and/or loop diuretics, antiepileptics) during the study
* Planned excessive exposure of area(s) to be treated with study medication to either natural or artificial sunlight (including tanning booths, sunlamps etc.) during the study
* Oestrogen therapy (including contraceptives), antidepressant medications and any other medication known to affect cortisol levels or HPA axis integrity within 4 weeks prior to SV2
* Cytochrome P450 3A4 (CYP 3A4) inducers (e.g., barbiturates, phenytoin, rifampicin) within 4 weeks prior to SV2
* Systemic cytochrome P450 3A4 (CYP 3A4) inhibitors (e.g., ketoconazole, itraconazole, metronidazole) within 4 weeks prior to SV2
* Topical cytochrome P450 3A4 (CYP 3A4) inhibitors (e.g., ketoconazole) within 2 weeks prior to SV2
* Non-nocturnal sleep patterns (e.g. night shift workers)
* Any of the following conditions, whether known or suspected:

  * depression and endocrine disorders (e.g. Cushing's disease, Addison's disease, diabetes mellitus) known to affect cortisol levels or HPA axis integrity
  * disorders of calcium metabolism associated with hypercalcaemia
  * cardiac disorders associated with abnormal QT intervals or rhythm disturbances including clinically significant bradycardia or tachycardia
  * severe renal insufficiency
  * severe hepatic disorders
* Any clinically significant abnormality following blood pressure/heart rate measurement or review of screening laboratory tests (blood and spot urine samples) collected at SV2
* Any clinically significant abnormality following physical examination at SV1
* Current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis
* Any of the following conditions present on the study treatment areas (trunk, limbs and scalp): viral (e.g., herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, ulcers and wounds
* Other inflammatory skin disorders (e.g. seborrhoeic dermatitis and contact dermatitis) that may confound the evaluation of psoriasis vulgaris
* Current participation in any other interventional clinical trial
* Previously enrolled in this trial
* Known or suspected of not being able to comply with the trial protocol (e.g., alcoholism, drug dependency or psychotic state)
* Females who are pregnant, wishing to become pregnant during the study or who are breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Taraska, Principal Investigator — Winnipeg Clinic
Locations (10):
- Canada (10):
  - Guildford Dermatology Specialists, Surrey, British Columbia
  - PerCuro Clinical Research, Victoria, British Columbia
  - Winnipeg Clinic Dermatology Research, Winnipeg, Manitoba
  - Maritime Medical Research Center, Bathurst, New Brunswick
  - Ultranova Skincare, Barrie, Ontario
  - Co-Medica, Courtice, Ontario
  - Mediprobe Research, London, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Centre de Dermatologie Maizerets, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Taraska V, Tuppal R, Olesen M, Bang Pedersen C, Papp K. Fixed combination aerosol foam calcipotriene (Cal) 0.005% plus betamethasone 0.064% (as dipropionate; BD) exhibits no impact on the HPA axis and calcium homeostasis in patients with extensive psoriasis vulgaris: a multicenter, single-arm, Phase II, 4-week MUSE study. Semin Cutan Med Surg. 2015;34 S1:PA-29.
- [Result] Taraska V, Tuppal R, Olesen M, Bang Pedersen C, Papp K. Fixed combination aerosol foam calcipotriene 0.005% (Cal) plus betamethasone dipropionate 0.064% (BD) exhibits no impact on the HPA axis and calcium homeostasis in patients with extensive psoriasis vulgaris: a multicenter, single-arm, Phase II, 4-week MUSE study. Semin Cutan Med Surg 2014;33:abst PA-13.
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit: 4-Jun-2012 Last Subject Last Visit: 2-May-2013
Pre-assignment Details: Subjects with extensive psoriasis vulgaris of at least moderate severity (according to the Investigators Global Assessment of Disease Severity; IGA) on the trunk, limbs and the scalp were enrolled.
  Screening: normal HPA axis function before and after ACTH-challenge test and albumin-corrected serum Ca lvl below the upper normal limit were required.
Groups:
- LEO 90100: LEO 90100: Calcipotriol 50 mcg/g (as hydrate) and betamethasone 0.5 mg/g (as dipropionate) Once daily for up to 4 weeks
Period: Overall Study
Arm/Group | LEO 90100
Started | 37
Completed | 35
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Serum Cortisol Concentration of ≤18 mcg/dl at 30 Minutes After Adrenocorticotrophic Hormone-challenge (ACTH-challenge)
Description: HPA-axis testing by means of the rapid standard-dose cosyntropin test (ACTH-challenge test) for detection of adrenal suppression.
Time Frame: Day 28
Population: Per protocol analysis set.
Measure: Number; unit: Subjects
Arm/Group | LEO 90100
Number analyzed (Participants) | 35
Subjects | 0

2. Primary Outcome: Change in Albumin-corrected Serum Calcium From Baseline to Day 28
Description: The effect of LEO 90100 on calcium metabolism was evaluated based on change in albumin-corrected serum calcium from Baseline to Day 28.
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
mmol/L | 0.014 (0.202)

3. Primary Outcome: Change in 24-hour Urinary Calcium Excretion From Baseline to Day 28
Description: The effect of LEO 90100 on calcium metabolism was evaluated based on change in 24-hour urinary calcium excretion from Baseline to Day 28 in 24-hour.
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: mmol/24H
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
mmol/24H | -0.49 (1.37)

4. Primary Outcome: Change in 24-hour Urinary Calcium:Creatinine Ratio From Baseline to Day 28
Description: The effect of LEO 90100 on calcium metabolism was evaluated based on change in urinary calcium:creatinine ratio from Baseline to Day 28.
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
mmol/g | -0.0300 (1.3997)

5. Secondary Outcome: Number of Subjects With Serum Cortisol Concentration of ≤18 mcg/dl at 30 and 60 Minutes After ACTH-challenge at Day 28
Description: Serum cortisol concentrations at 30 and 60 minutes after injection were measured in order to assess the maximum stimulated cortisol level achieved. Potential adrenal suppression was indicated if the serum cortisol concentration is ≤18mcg/dl at 30 minutes after the injection.
Time Frame: Day 28
Measure: Number; unit: Subjects
Arm/Group | LEO 90100
Number analyzed (Participants) | 35
Subjects | 0

6. Secondary Outcome: Number of Participants With an Adverse Drug Reaction (ADR)
Description: Adverse drug reactions (ADRs) were defined as adverse events for which the investigator has not described the causal relationship to investigational medication as "not related".
Time Frame: Baseline to Day 28
Measure: Number; unit: participants
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
participants | 1

7. Secondary Outcome: Change in Serum Phosphate From Baseline to Day 28
Description: The effect of LEO 90100 on calcium metabolism was evaluated based on change in serum phosphate from Baseline to Day 28.
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
mmol/L | 0.030 (0.145)

8. Secondary Outcome: Change in 24-hour Urinary Phosphate Excretion From Baseline to Day 28
Description: The effect of LEO 90100 on calcium metabolism was evaluated based on change in 24-hour urinary phosphate excretion from Baseline to Day 28.
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: mmol/24H
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
mmol/24H | -0.25 (8.67)

9. Secondary Outcome: Change in Urinary Phosphate: Creatinine Ratio From Baseline to Day 28
Description: The effect of LEO 90100 on calcium metabolism was evaluated based on change in urinary phosphate:creatinine ratio from Baseline to Day 28.
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
mmol/g | 1.847 (6.215)

10. Secondary Outcome: Change in Serum Alkaline Phosphatase (ALP) From Baseline to Day 28
Description: The effect of LEO 90100 on calcium metabolism was evaluated based on change in serum ALP from Baseline to Day 28.
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
IU/L | -1.5 (12.5)

11. Secondary Outcome: Change in Plasma Parathyroid Hormone (PTH) From Baseline to Day 28
Description: The effect of LEO 90100 on calcium metabolism was evaluated based on change in plasma PTH from Baseline to Day 28.
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
pmol/L | 0.893 (2.207)

12. Secondary Outcome: Change in Blood Pressure From Baseline to Day 28
Description: The effect of LEO 90100 on calcium metabolism was evaluated based on vital sign assessments (blood pressure).
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
mmHg
  Diastolic Blood Pressure (mmHg) | -1.5 (6.2)
  Systolic Blood Pressure (mmHg) | -2.2 (8.1)

13. Secondary Outcome: Change in Heart Rate From Baseline to Day 28
Description: The effect of LEO 90100 on calcium metabolism was evaluated based on vital sign assessments (heart rate).
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
beats/min | 0.2 (10.4)

14. Secondary Outcome: Number of Subjects Who Discontinued From the Study
Description: Number of subjects who discontinued from the study due to adverse events.
Time Frame: Baseline to Day 28
Measure: Number; unit: participants
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
participants | 0

15. Secondary Outcome: Pharmacokinetic Evaluation Cmax
Description: The following PK parameters will be calculated, if possible, for each assayed compound based on the obtained plasma concentrations:
  * AUC0-t
  * AUC0-∞
  * Cmax
  * Tmax
  * T½
  If it is not possible to calculate the above PK parameters, samples with plasma concentration above lower limit of quantification (LLOQ) will be presented.
  All subjects but 1 had plasma concentration of calcipotriol below the LLOQ (lower limit of quantification), and thus it was not possible to calculate group mean of the derived PK parameter based on one sample. Provided values for calcipotriol Cmax are derived from that 1 subject.
Time Frame: 4 weeks / 28 days
Population: Plasma samples for PK assessment were collected from all 37 subjects however; PK samples from 2 subjects were only collected at screening (SV2) and at Day 14. Therefore these 2 subjects were excluded from PK analysis. Summary of PK parameters based on those subjects that had quantifiable plasma concentrations.
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | LEO 90100
Number analyzed (Participants) | 35
pg/ml
  Betamethasone dipropionate (BDP) (n=5) | 52.2 [33.7 to 81.1]
  betamethasone 17- propionate (n=27) | 148 [30.2 to 1133]
  calcipotriol (n=1) | 55.9 [55.9 to 55.9]
  MC1080 (n=5) | 24.4 [23.3 to 26.6]

16. Secondary Outcome: Pharmacokinetic Evaluation AUClast
Description: The following PK parameters will be calculated, if possible, for each assayed compound based on the obtained plasma concentrations:
  * AUC0-t
  * AUC0-∞
  * Cmax
  * Tmax
  * T½
  If it is not possible to calculate the above PK parameters, samples with plasma concentration above lower limit of quantification (LLOQ) will be presented.
  All subjects but 1 had plasma concentration of calcipotriol below the LLOQ (lower limit of quantification), and thus it was not possible to calculate group mean of the derived PK parameter based on one sample. Provided values for calcipotriol AUClast are derived from that 1 subject.
Time Frame: 4 weeks / 28 days
Population: as for outcome 15
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | LEO 90100
Number analyzed (Participants) | 35
pg/ml
  Betamethasone dipropionate (BDP) (n=5) | 36.5 [16.9 to 82.5]
  betamethasone 17- propionate (n=27) | 683.6 [18.5 to 4254]
  calcipotriol (n=1) | 82.5 [82.5 to 82.5]
  MC1080 (n=5) | 59.3 [55.3 to 65.5]

17. Secondary Outcome: Pharmacokinetic Evaluation AUCinf
Description: The following PK parameters will be calculated, if possible, for each assayed compound based on the obtained plasma concentrations:
  * AUC0-t
  * AUC0-∞
  * Cmax
  * Tmax
  * T½
  If it is not possible to calculate the above PK parameters, samples with plasma concentration above lower limit of quantification (LLOQ) will be presented.
Time Frame: 4 weeks / 28 days
Population: as for outcome 15
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | LEO 90100
Number analyzed (Participants) | 35
pg/ml
  Betamethasone dipropionate (BDP) (n=5) | NA [NA to NA] — It was not possible to estimate λz (elimination phase rate constant) to calculate AUCinf for any of the 4 analytes after use of LEO 90100 (assay sensitivity limitations, insufficient plasma concentration data in the terminal phase of PK curves).
  betamethasone 17- propionate (n=27) | NA [NA to NA] — It was not possible to estimate λz (elimination phase rate constant) to calculate AUCinf for any of the 4 analytes after use of LEO 90100 (assay sensitivity limitations, insufficient plasma concentration data in the terminal phase of PK curves).
  calcipotriol (n=1) | NA [NA to NA] — It was not possible to estimate λz (elimination phase rate constant) to calculate AUCinf for any of the 4 analytes after use of LEO 90100 (assay sensitivity limitations, insufficient plasma concentration data in the terminal phase of PK curves).
  MC1080 (n=5) | NA [NA to NA] — It was not possible to estimate λz (elimination phase rate constant) to calculate AUCinf for any of the 4 analytes after use of LEO 90100 (assay sensitivity limitations, insufficient plasma concentration data in the terminal phase of PK curves).

18. Secondary Outcome: Pharmacokinetic Evaluation Tmax
Description: The following PK parameters will be calculated, if possible, for each assayed compound based on the obtained plasma concentrations:
  * AUC0-t
  * AUC0-∞
  * Cmax
  * Tmax
  * T½
  If it is not possible to calculate the above PK parameters, samples with plasma concentration above lower limit of quantification (LLOQ) will be presented.
  All subjects but 1 had plasma concentration of calcipotriol below the LLOQ (lower limit of quantification), and thus it was not possible to calculate group mean of the derived PK parameter based on one sample. Provided values for calcipotriol Tmax are derived from that 1 subject.
Time Frame: 4 weeks / 28 days
Population: as for outcome 15
Measure: Median (Full Range); unit: h
Arm/Group | LEO 90100
Number analyzed (Participants) | 35
h
  Betamethasone dipropionate (BDP) (n=5) | 1.0000 [1.000 to 3.050]
  betamethasone 17- propionate (n=27) | 2.0830 [0.00 to 7.05]
  calcipotriol (n=1) | 2.000 [2.000 to 2.000]
  MC1080 (n=5) | 5.0000 [3.000 to 5.000]

19. Secondary Outcome: Pharmacokinetic Evaluation T1/2
Description: as for outcome 17
Time Frame: 4 weeks / 28 days
Population: as for outcome 15
Measure: Mean (Full Range); unit: h
Arm/Group | LEO 90100
Number analyzed (Participants) | 35
h
  Betamethasone dipropionate (BDP) (n=5) | NA [NA to NA] — It was not possible to estimate λz (elimination phase rate constant) to calculate T1/2 for any of the 4 analytes after use of LEO 90100 (assay sensitivity limitations, insufficient plasma concentration data in the terminal phase of PK curves).
  betamethasone 17- propionate (n=27) | NA [NA to NA] — It was not possible to estimate λz (elimination phase rate constant) to calculate T1/2 for any of the 4 analytes after use of LEO 90100 (assay sensitivity limitations, insufficient plasma concentration data in the terminal phase of PK curves).
  calcipotriol (n=1) | NA [NA to NA] — It was not possible to estimate λz (elimination phase rate constant) to calculate T1/2 for any of the 4 analytes after use of LEO 90100 (assay sensitivity limitations, insufficient plasma concentration data in the terminal phase of PK curves).
  MC1080 (n=5) | NA [NA to NA] — It was not possible to estimate λz (elimination phase rate constant) to calculate T1/2 for any of the 4 analytes after use of LEO 90100 (assay sensitivity limitations, insufficient plasma concentration data in the terminal phase of PK curves).

20. Secondary Outcome: Efficacy Evaluation
Description: The percentage of subjects who achieved 'controlled disease' (i.e., Clear or Almost clear) according to the Investigator's Global Assessment (IGA) of disease severity on the trunk, limbs and scalp at Days 28 (Visit 3) and End of treatment (EoT) were presented.
Time Frame: 4 weeks I 28 days and End of treatment
Population: The percentage of subjects achieving controlled disease on Day 28 (n=35) was calculated from the full analysis set.
  The percentage of subjects achieving controlled disease at End of Treatment (n=37) was was calculated from the full analysis set using a last observation carried forward approach.
Measure: Number; unit: percentage of subjects
Arm/Group | LEO 90100
Number analyzed (Participants) | 37
percentage of subjects
  Day 28 (n=35) | 48.6
  End of treatment (n=37) | 45.9

ADVERSE EVENTS:
Arm/Group | LEO 90100
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 4/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 90100 (N=37)
Fungal infection (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — considered by the Investigator to be probably related to treatment (an adverse drug reaction (ADR))

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.